CLINICAL TRIAL: NCT00054535
Title: Treatment Of Patients With Metastatic Melanoma Using Recombinant Vaccinia And Fowlpox Viruses Encoding The Tyrosine Antigen In Combination With Interleukin-2
Brief Title: Vaccine Therapy and Interleukin-2 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000270794; NCI-03-C-0080; NCI-6119; NCT00051610 (obsolete NCT alias)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2004-07

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant fowlpox-tyrosinase vaccine
Biological: vaccinia-tyrosinase vaccine

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response that will kill tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill melanoma cells.

PURPOSE: Phase II trial to study the effectiveness of combining vaccine therapy with interleukin-2 in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate (partial response or complete remission) in patients with metastatic melanoma treated with vaccinia-tyrosinase vaccine, fowlpox-tyrosinase vaccine, and high-dose interleukin-2.
* Determine the immunologic response, measured by the reactivity of CD4+ and CD8+ T cells and serum immunoglobulins against tyrosinase and melanoma cells, in patients treated with this regimen.

OUTLINE: Patients receive vaccinia-tyrosinase vaccine intramuscularly (IM) on day 1 followed by fowlpox-tyrosinase vaccine IM on days 15 and 29. Patients then receive high-dose interleukin-2 (IL-2) IV over 15 minutes every 8 hours beginning on day 30 for up to 12 doses and again beginning approximately 3 weeks after the initial dose. Patients with stable disease or a minor, mixed, or partial response may receive additional courses of fowlpox-tyrosinase vaccine (2 doses) and IL-2 as above in the absence of disease progression or unacceptable toxicity. Patients with a complete response (CR) receive 1 additional course beyond achieving CR.

Patients are followed annually for at least 5 years.

PROJECTED ACCRUAL: A total of 19-35 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic melanoma

  * Measurable disease
  * Disease progression while receiving prior standard treatment
  * No ocular or mucosal primary site
* No uncontrolled brain metastases

PATIENT CHARACTERISTICS:

Age

* 16 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* WBC at least 3,000/mm^3
* Platelet count at least 90,000/mm^3
* No coagulation disorders

Hepatic

* Bilirubin no greater than 1.6 mg/dL (less than 3.0 mg/dL in patients with Gilbert's syndrome)
* AST/ALT less than 3 times normal
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal

* Creatinine no greater than 1.6 mg/dL

Cardiovascular

* No major cardiovascular illness

Pulmonary

* No major respiratory illness

Immunologic

* HIV negative
* No autoimmune disease
* No active systemic infections
* No primary or secondary immunodeficiency (e.g., hereditary disorders such as ataxia-telangiectasia or Wiskott-Aldrich syndrome or acquired immunodeficiencies after bone marrow transplantation)
* No allergy to eggs
* No prior allergy or untoward reaction to smallpox vaccination (if previously vaccinated)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No close contact with the following individuals for 2 weeks after vaccinia vaccination:

  * Children under 5 years of age
  * Pregnant women
  * Individuals with prior or active eczema or other eczematoid skin disorders
  * Individuals with other acute, chronic, or exfoliative skin conditions (e.g., burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds)
  * Immunosuppressed individuals
* No active atopic dermatitis
* No prior or active eczema
* No active cases of the following conditions:

  * Extensive psoriasis
  * Severe acneiform rash
  * Impetigo
  * Varicella zoster
  * Burns
  * Traumatic or pruritic skin conditions
  * Open wounds
* No unhealed surgical scars

  * Healed surgical stomas (e.g., colostomy) allowed

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior recombinant vaccinia or fowlpox vaccines for melanoma
* No prior vaccination with full length tyrosinase protein, or a vector encoding the full length protein for melanoma

  * Prior individual tyrosinase peptides are allowed
* No prior high-dose interleukin-2

Chemotherapy

* Not specified

Endocrine therapy

* No concurrent oral, IV, topical, or inhaled steroids

Radiotherapy

* Not specified

Surgery

* Recovered from prior surgery

Other

* Recovered from prior therapy for melanoma
* More than 3 weeks since prior systemic therapy for melanoma
* No other concurrent systemic therapy for melanoma

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-01; Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne L. Topalian, MD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States